CLINICAL TRIAL: NCT01437618
Title: FOLFOXIRI Plus Bevacizumab as First-line Treatment for BRAF V600E Mutant Metastatic Colorectal Cancer: a Prospective Evaluation
Brief Title: First-line FOLFOXIRI Plus Bevacizumab in BRAF Mutant Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Alfredo Falcone, Professor Alfredo Falcone, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: BRAF-0809-TRIBV
Record Dates: First submitted 2011-07-12; First posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- BRAF mutant mCRC
  Interventions: Drug: FOLFOXIRI plus bevacizumab

INTERVENTIONS:
Drug: FOLFOXIRI plus bevacizumab — * BEVACIZUMAB 5 mg/Kg i.v. over 30', day 1 followed by
  * IRINOTECAN 165 mg/sqm i.v. over 1-h, day 1 followed by
  * OXALIPLATIN 85 mg/sqm i.v. over 2-h, day 1 concomitantly with
  * l-LV 200 mg/sqm i.v. over 2-h, day 1 followed by
  * 5-FLUOROURACIL 3200 mg/sqm i.v. 48-h continuous infusion, starting on day 1 Cycles repeated every 2 weeks

SUMMARY:
The purpose of this study is to prospectively verify if FOLFOXIRI plus bevacizumab as first-line treatment could be considered a promising approach to improve the outcome of BRAF mutant metastatic colorectal cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma;
* Availability of formalin-fixed paraffin embedded tumor block from primary and/or metastasis;
* BRAF V600E mutant status of primary colorectal cancer and/or related metastasis;
* Unresectable and measurable metastatic disease according to RECIST criteria;
* Male or female, aged > 18 years and < 75 years;
* ECOG PS < 2 if aged < 71 years;
* ECOG PS = 0 if aged 71-75 years;
* Life expectancy of more than 3 months;
* Adequate haematological function: ANC ≥ 1.5 x 10^9/L; platelets ≥ 100 x 10^9/L, Hb ≥ 9 g/dL;
* Adequate liver function: serum bilirubin ≤ 1.5 x ULN; alkaline phosphatase and transaminases ≤ 2.5 x ULN (in case of liver metastases ≤ 5 x ULN);
* Serum creatinine ≤ 1.5 x ULN;
* Previous adjuvant chemotherapy is allowed if more than 12 months have elapsed between the end of adjuvant therapy and first relapse;
* At least 6 weeks from prior extended radiotherapy and 4 weeks from surgery;
* Written informed consent to experimental treatment and molecular analyses.

Exclusion Criteria:

* Presence or history of CNS metastasis;
* Serious, non-healing wound, ulcer, or bone fracture;
* Evidence of bleeding diathesis or coagulopathy;
* Uncontrolled hypertension;
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (CVA) (≤6 months before treatment start), myocardial infarction (≤ 6 months before treatment start), unstable angina, NYHA ≥ grade 2 chronic heart failure (CHF), uncontrolled arrhythmia;
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes;
* Chronic, daily treatment with high-dose aspirin (>325 mg/day);
* Symptomatic peripheral neuropathy ≥ 2 grade NCIC-CTG criteria;
* Active uncontrolled infections;
* Treatment with any investigational drug within 30 days prior to enrolment;
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of curatively treated basal and squamous cell carcinoma of the skin or in situ cancer of the cervix;
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start;
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome;
* Fertile women (< 2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BRAF mutant mCRC
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-06; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | About 24-30 months (From treatment initiation to evidence of progression or death from any cause)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, Italy

REFERENCES:
- [Derived] Loupakis F, Cremolini C, Salvatore L, Masi G, Sensi E, Schirripa M, Michelucci A, Pfanner E, Brunetti I, Lupi C, Antoniotti C, Bergamo F, Lonardi S, Zagonel V, Simi P, Fontanini G, Falcone A. FOLFOXIRI plus bevacizumab as first-line treatment in BRAF mutant metastatic colorectal cancer. Eur J Cancer. 2014 Jan;50(1):57-63. doi: 10.1016/j.ejca.2013.08.024. Epub 2013 Oct 15. PMID 24138831